CLINICAL TRIAL: NCT04147182
Title: Perioperative Intravesical Instilation of Hypertonic Saline Following Bladder
Brief Title: Perioperative Intravesical Instilation of Hypertonic Saline Following Bladder Tumor Resection
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dan Leibovici (Other)
Responsible Party: Sponsor-Investigator, Dan Leibovici, Professor Dan Leibovici- Head of the Urology department of Kaplan MC, Kaplan Medical Center
Organization: Kaplan Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0116-17-KMC
Record Dates: First submitted 2019-10-23; First posted 2019-10-31 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: TCC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient with low grade TCC (Experimental): 1. Patients of 18 years or older able to sign informed consent
  2. A previous diagnosis of low grade bladder cancer
  3. A pyelographic imaging examination (CTU, MRU, IVP, antegrade/retrograde pyelography) showing normal upper urinary tract in the 12 months prior to inclusion
  4. Serum creatinine levels ≤ 2.0 mg/dl
  5. Serum sodium levels <146 mg/ml
  6. Current bladder tumor diagnosed by endoscopy or imaging in the last 3 months
  7. Patient is candidate for TURBT
  Interventions: Drug: Hypertonic Saline 3%

INTERVENTIONS:
Drug: Hypertonic Saline 3% — 3% and 5% Sodium Chloride Injection, USP is a sterile, nonpyrogenic, hypertonic solution for fluid and electrolyte replenishment in single dose containers for intravenous administration. The pH may have been adjusted with hydrochloric acid. It contains no antimicrobial agents.

SUMMARY:
Hypertonic saline at the concentration of 3% (hypersel) has been injected for years into echinococcal cysts to kill live scolices, and is also known to kill suspended cells by means of a steep osmotic gradient and the investigators postulate that perioperative intravesical instillation of hypersel for patients with low grade bladder cancer is safe and may be active against shedded and suspended tumor cells and thus may decrease recurrence risk.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of 18 years or older able to sign informed consent
2. A previous diagnosis of low grade bladder cancer
3. A pyelographic imaging examination (CTU, MRU, IVP, antegrade/retrograde pyelography) showing normal upper urinary tract in the 12 months prior to inclusion
4. Serum creatinine levels ≤ 2.0 mg/dl
5. Serum sodium levels <146 mg/ml
6. Current bladder tumor diagnosed by endoscopy or imaging in the last 3 months
7. Patient is candidate for TURBT

Exclusion Criteria:

1. Previous history of high grade bladder cancer including carcinoma in situ
2. Presence of upper urinary tract tumor on imaging
3. Renal failure with serum creatinine >2.0 mg/dl prior to inclusion
4. Hypernatremia >146 mg/dl prior to inclusion
5. Contra-indication to undergo TURBT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-12-02 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2020-11-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as assessed by Common Terminology Criteriafor Adverse Events of Renal and urinary disorders (CTCAE)Version 5.0,2017, Satisfaction assessed by Clavien-Dindo. | 12 month
  The investigators monitored the Sodium levels in the blood after the administration of the Hypertonic Saline and documented and measure side effects by Clavien-Dindo scale

CONTACTS AND LOCATIONS:
Locations (1):
- Kaplan MC, Rehovot, Israel

IPD SHARING:
Plan to Share IPD: No